CLINICAL TRIAL: NCT06230497
Title: Correlation Analysis Between Mostcare Parameters and Spontaneous Breathing Trial in Patients After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 216-4
Record Dates: First submitted 2024-01-17; First posted 2024-01-30 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-03

CONDITIONS: Post-cardiac Surgery; Ventilator Weaning
Keywords: Post-cardiac Surgery; Ventilator weaning; Mostcare; ressure recording analytical method

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac output (CO) monitoring is of primary importance in high-risk surgery and critically ill patients.

Intermittent thermodilution (ThD) by means of a pulmonary artery catheter (PAC) was invasiveness, the occurrence of complications, and inability to estimate CO on a beat-by-beat basis may explain the reduction in routine use. Echocardiography is now widely used. However, a poor acoustic window, inaccurate diameter calculations, and difficulty maintaining the angle of insonation and blood flow within the recommended values may lead to inaccuracy in CO estimation.Pulse contour methods (PCMs) are commonly used as they seem to fulfill most of the characteristics of an "ideal" hemodynamic monitoring system.

Mostcare can continuously and real-time monitor important circulatory indicators such as cardiac output, peripheral vascular resistance index (SVRI), cardiovascular impedance (Ztot), cardiac cycle efficiency (CCE), and maximum pressure gradient (dp/dt MAX). It may help identify the causes of difficulty in weaning patients from ventilators after cardiac surgery.

DETAILED DESCRIPTION:
Cardiac output (CO) monitoring is of primary importance in high-risk surgery and critically ill patients.

Intermittent thermodilution (ThD) by means of a pulmonary artery catheter (PAC) has been used as the reference method and to validate alternative monitoring systems. Its invasiveness, the occurrence of complications, and inability to estimate CO on a beat-by-beat basis may explain the reduction in routine use.

Echocardiography is now widely used in ICUs for the complete assessment of heart function, volume status, and CO measurement. Because it has been well accepted as a first-line diagnostic tool for circulatory failure, it has been proposed as an alternative for ThD to evaluate CO in selected patient populations . A poor acoustic window, inaccurate diameter calculations, and difficulty maintaining the angle of insonation and blood flow within the recommended values may lead to inaccuracy in CO estimation.Finally, training is of major importance.

Pulse contour methods (PCMs) are commonly used in operating rooms or ICUs as they seem to fulfill most of the characteristics of an "ideal" hemodynamic monitoring system.

Mostcare can continuously and real-time monitor important circulatory indicators such as cardiac output, peripheral vascular resistance index (SVRI), cardiovascular impedance (Ztot), cardiac cycle efficiency (CCE), and maximum pressure gradient (dp/dt MAX). It may help identify the causes of difficulty in weaning patients from ventilators after cardiac surgery.

This is a prospective observational study. Patients admitted to the ICU after cardiac surgery and mechanically ventilated for more than 24 hours were monitored for mostcare before attempting to withdraw from the ventilator, and assessment of systemic circulation and cardiac ultrasound was completed.

Patients were given an spontaneous breathing test(SBT) off the ventilator. Mostcare parameters were also recorded. If the SBT experiment was successful the endotracheal tube was removed, if it failed then mostcare monitoring and assessment of circulation and ultrasound were performed again after resumption of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the ICU after cardiac surgery
2. mechanically ventilated for more than 24 hours

Exclusion Criteria:

1. the presence of pathologies that could affect the quality and reliability of the arterial pulse transmission (aortic valve diseases, aortic aneurysm or dissection, thoracic outlet syndrome);
2. arrhythmias;
3. hemodynamic instability;
4. age less than 18 years or more than 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU after cardiac surgery and mechanically ventilated for more than 24 hours
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
The Cardiac Cycle Efficiency (CCE)(unit) | Day1
  The Cardiac Cycle Efficiency (CCE) parameter provided by Mostcare is a comprehensive index of cardiac function that takes into account the mechanical and geometric properties of the heart. It integrates the changes in pressure and volume throughout the cardiac cycle to provide a single value that reflects the heart's efficiency.
  CCE is computed as CCE= Wsys/Wbeat*K(t), where Wsys is the power function from the systolic pressure wave, Wbeat is the power function from the entire cardiac cycle pressure wave, and K(t) is the ratio of mean pressure expected over mean pressure measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine of pekin union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided